CLINICAL TRIAL: NCT02288871
Title: Pilot Trial: Comparison of Flow Patterns. Is There a Difference Between sewed-in and "Sutureless" Bioprosthetic Aortic Heart Valves?
Brief Title: Pilot Trial: Comparison of Flow Patterns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Alfred A Kocher, MD, Professor, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1790/2013-1
Record Dates: First submitted 2014-10-22; First posted 2014-11-11 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: aortic valve replacement; aortic valve bioprosthesis; hemodynamics
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

ARMS (2):
- "Sutureless" valve (Other): Patients who underwent aortic valve replacement with a "sutureless" aortic valve.
  An echocardiogram and a cardiac CT-scan will be conducted.
  Interventions: Radiation: Cardiac CT-scan
- "Sewed-in" valve (Other): Patients who underwent aortic valve replacement with a "sewed-in" aortic valve. An echocardiogram and a cardiac CT-scan will be conducted.
  Interventions: Radiation: Cardiac CT-scan

INTERVENTIONS:
Radiation: Cardiac CT-scan — ECG gated CT angiography of the heart will be performed on a 128-slice dual-source and two Stellar detectors CT system with retrospective ECG-gating (Siemens/SOMATOM Definition Flash - Siemens, Germany, 100kV, 395.75 mAs).
  In details, multi-phase images will be acquired to reconstruct between 10 and 100% of the cardiac cycle (10% increments) with a slice thickness of 1 mm. Examination will include left ventricular outflow tract, aortic root, coronary sinus, ascending aorta together with the prosthetic valves.

SUMMARY:
The purpose of this study is to determine why sutureless aortic bioprostheses apparently offer better haemodynamic properties compared to sewed-in aortic bioprostheses in patients who underwent aortic valve replacement.

Our approach to address this question is the combination of clinical data with the application of specifically validated experimental and computer based analyses to compare the performance of these valves under patient-specific conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent open aortic valve replacement with either an Edwards Magna Ease or an Edwards Intuity valve
* Implanted valve size 23mm
* Surgical access via full sternotomy or hemisternotomy
* Intuity Valve System implanted by one of the clinical investigators of the TRITON trial (http://clinicaltrials.gov/show/NCT01445171) at the Medical University of Vienna
* Post-operative ejection fraction ≥50%
* Sinus-Rhythm
* Ability to understand and comply with study procedures
* Signed informed consent

Exclusion Criteria:

* Under 18 years of age
* Emergency surgery
* Pregnancy
* Previous aortic root replacement
* Previous aortic valve replacement
* Previous or concomitant root enlargement
* Previous or concomitant repair of the ascending aorta
* Paravalvular leakage
* Ectasia of the ascending aorta
* Previous or concomitant myomectomy
* Concomitant replacement or repair of valves other than aortic
* Usage of more than 3 sutures for implantation of the Intuity Valve System
* Heavily calcified aortic root
* Glomerular filtration rate (GFR) < 30 ml/min
* Inability to understand or comply with study procedures
* Known allergic reaction to iodinated, non-ionic contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of maximum and minimum velocity under patient specific conditions | between 6 months and 4 years after aortic valve replacement
Comparison of the effective orifice area under patient specific conditions | between 6 months and 4 years after aortic valve replacement
Comparison of the percentage of turbulent flow under patient specific conditions | between 6 months and 4 years after aortic valve replacement
Comparison of the pressure drop under patient specific conditions | between 6 months and 4 years after aortic valve replacement

SECONDARY OUTCOMES:
Patient-specific, computer simulated pressure gradients compared to echocardiographically obtained pressure gradients. | between 6 months and 4 years after aortic valve replacement
  The first secondary outcome measure is the comparison of
  -pressure gradients
  as computed by the model against the same data collected standardly with echocardiographic technique. Differences will be quantified.
  If positive (< 10%), this assessment would enhance the use of patient-specific models in clinics as a predictive tool for detailed haemodynamics."
Patient-specific, computer simulated peak velocity compared to echocardiographically obtained peak velocity. | between 6 months and 4 years after aortic valve replacement
  The second secondary outcome measure is the comparison of
  -peak velocity
  as computed by the model against the same data collected standardly with echocardiographic technique. Differences will be quantified.
  If positive (< 10%), this assessment would enhance the use of patient-specific models in clinics as a predictive tool for detailed haemodynamics."

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Kocher, MD, Principal Investigator — Division of Cardiac Surgery, Department of Surgery, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria